CLINICAL TRIAL: NCT05546073
Title: Advanced Use of Point-of-care Technology Versus Usual Care During In-home-assessment by Acute Community Nurses in Older Adults for Reducing Acute Hospital Admissions
Brief Title: Advanced Point-of-care Technology During In-home Assessment Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense Patient Data Explorative Network (Other); Region of Southern Denmark (Other); Kolding Municipality, Denmark (Unknown); Karen Elise Jensen Foundation (Other); AP Moeller Foundation (Other); Hartmann Fonden (Other); Merchant L. F. Foghts Foundation (Unknown); Director Emil C Hertz and wife Inger Hertz Foundation (Unknown); Gangsted Foundation (Unknown); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20220050
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Acute Respiratory Disease; Acute Illness
Keywords: acute illness; older adults; acute home care; pre-hospital care; point-of-care technology; geriatric; acute community nurse; focused lung ultrasound scan; FLUS

STUDY DESIGN:
Intervention Model Description: 632 participants referred to the acute community health care service for in-home assessment due to acute disease will be enrolled and randomized 1:1 to receive usual care or advanced point-of-care technology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Usual Care (No Intervention): Participants in the control-arm will undergo usual care. This covers clinical inspection, vital parameters (respiratory rate(breaths/min), saturation (%), blood pressure (mmHg), heart rate (beats/min), body temperature (celsius), and Glasgow Coma Scale) , and point-of-care blood-test for CRP and haemoglobin
- Intervention - Advanced point-of-care technology (Experimental): Participants in the intervention-arm will undergo usual care as well as advanced point-of-care technology.
  Interventions: Other: Advanced point-of-care technology

INTERVENTIONS:
Other: Advanced point-of-care technology — The intervention consists of:
  * focused lung ultrasound scan(FLUS)
  * venous blood samples for leucocytes with 5-part differential count, creatinin, sodium, potassium, urea
  Arms: Intervention - Advanced point-of-care technology

SUMMARY:
Due to ageing-related physiological changes, diagnosing older adults is challenging. Delayed disease recognition lead to adverse health outcomes and increased hospitalisation, which is why there is a need to develop new procedures for timely diagnosis and treatment of older adults. Point-of-care technology, e.g. focused lung ultrasound scan and bedside analysis of blood samples (leucocytes with differential count, electrolytes and creatinine) carried out in the patients' home may support clinical decision-making, and potentially reduce acute hospital admissions.

The trial's overall aim is to investigate whether increased point-of-care technology, i.e. focused lung ultrasound scan and bedside blood analysis, used as in-home diagnostics in older adults with acute respiratory symptoms, can qualify the general practitioner's clinical decision-making for early treatment initiation and eventually reduce acute hospital admission.

DETAILED DESCRIPTION:
The trial is conducted in Kolding municipality in Denmark. Participants eligible for this study are people aged 65 years or older, referred to the Acute Community Health Care Service (ACHCS) in Kolding municipality for an in-home assessment.

Data collection:

In the control group, the Acute Community Nurses (ANC) will carry out usual care that involves a clinical inspection, measurements of vital signs (respiratory rate(breaths/min), saturation (%), blood pressure (mmHg), heart rate (beats/min), body temperature (celsius), and Glasgow Coma Scale), and point-of-care tests (POCT) for C-reactive protein (CRP) and haemoglobin.

In the intervention group, the ACN will carry out extended POCT besides usual care. Extended POCT covers a focused lung ultrasound scan (FLUS) and biochemical blood analyses. FLUS examination follows a standardized protocol (21). Biochemical analyses include sodium, potassium, creatinine, urea, and leucocytes with differential count.

In both control and intervention groups the ACN communicates the examination results to the participants' primary care physician (PCP) by telephone as well as an electronic written documentation. The findings will support the PCP in the clinical decision-making. The communication to the PCP is part of the usual care and is carried out in both groups.

Training of ACNs:

Prior to the study initiation, all ACNs are trained in FLUS examination, technical procedure of POCT biochemical blood-analysis, as well as in research methods with specific focus on study procedures to increase their adherence to and respect for to the randomization procedure and protocol.

Point-of-care technology used in the study:

FLUS is carried out using Lumify® C5-2 Curved Array Transducer (Philips Medical Systems, Bothell, WA), with a bandwidth of 5-2 megahertz (MHz) and scan depth up to 30 cm.

POCT on blood samples for creatinine and electrolytes are carried out using venous blood samples (collected in lithium/heparin vacutainers) and analysed immediately on the POCT instrument i-STAT® (Abbott, Inc., NJ, U.S.A.) using CHEM8 cassette.

POCT blood analysis for leucocyte differential count is carried out using venous blood samples (collected in EDTA-vacutainers) and analysed immediately on the POCT instrument HemoCue® WBF DIFF System (HemoCue AB, Ängelholm, Sweden) with dedicated micro-cuvettes.

POCT blood-analysis for CRP is carried out using blood samples obtained by finger-prick and analysed on the POCT instrument QuickRead go® (Orion Diagnostica, Oy).

Data-sources:

To assess co-morbidity, disabilities, utilization of primary care and health care services, death, and medical history external data sources will be applied for permission to access.

The Danish Health Data Authority is responsible for the national health registers containing data related to the health of the entire Danish population and services of the healthcare system. A unique personal identification number for all people living in Denmark makes it possible to link data across national health registers.

The Danish Health Data Authority will be applied to get access to the Danish National Patient Registry, the Danish Register of Causes of Death, The Danish National Prescription Registry, and the Danish National Health Service Register. The registers contain information about diseases, treatments, deaths, and health care utilization, and are needed to access information on comorbidity, time of death, medical history, treatment initiations or changes, and number of consultations at PCPs.

The Electronic Municipal Care Records (EOJ - Elektronisk Omsorgsjournal) registers the amount of home care the participants receive, and will be obtained at day 0 and at day 30 to investigate possible changes as a proxy of changes in functional level.

The hospital Electronic Patient Journal (EPJ) will be accessed by the primary investigator to register admissions, reason for admission and any complications during admission. The EPJ will be accessed at day 30 after the acute visit to register admissions, reasons for admission, length of admission, treatment during admission, functional decline during admission, and discharge diagnosis.

Data monitoring:

During the study, several checkpoints will be established to ensure adherence to protocol. Number of kits used will be noted every month to ensure no extra kits for POCT on biochemistry on blood samples are used as a violation to protocol. Time and date logging on each POCT device will be carried out each month to ensure adherence to protocol.

Sample size:

A clinically significant reduction of acute hospital admission is set to a 10% reduction. However, it is unknown how many patients are acutely admitted after the first visit of ACNs. Preliminary results from a pilot-study of the intervention (not yet published) showed that 21% of included participants were acutely admitted. We then assume to reduce hospital admissions by 10%, and to detect a reduction from 31% to 21% at a significance level 0.05 with a power of 80, a total of 602 participants are required (301 in each arm). Allowing for a 5 % drop out after randomisation, 316 in each arm are required (a total of 632 participants).

ELIGIBILITY:
Inclusion Criteria:

* referred to the ACHCS in Kolding Municipality for in-home assessment
* dyspnoea
* cough
* fever
* fall
* functional decline defined as either subjective (not able to perform normal daily activities as usual) or objective functional decline (increased need of home care)

Exclusion Criteria:

* moderate to severe cognitive impairment
* antibiotic treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 632 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Admission ≤ 30-days | 30 days
  Proportion of Admissions during 30 days follow-up

SECONDARY OUTCOMES:
Mortality ≤ 30-days | 30 days
  Proportion of diseased participants in the intervention group and control group after inclusion during 30 days follow-up
Acute admissions at day 0 | Day 0
  Proportion of acute admissions on visit day (day 0)
Length of hospital admission | 30 days
  Number of days admitted to acute-care hospital, long-term acute-care hospital or in an emergency department.
Hospital-free days ≤ 30-days | 30 days
  Number of days alive that is spend outside of an acute-care hospital, long-term acute-care hospital or in an emergency department, including days spent wholly or in part under "observation" status
Complications during hospital admission | 30 days
  Number of complications registered in the electronic patient journal during admission including delirium and fall
Treatment initiations or changes at day 0 | Day 0
  Number of treatment initiation or changed at day 0 including antibiotics, diuretics, inhalation medication, prednisolone, iv fluids, iv antibiotics
Treatment initiation or changes ≤ 30-day | 30 days
  Number of treatment initiation or changed during 30 days follow-up including antibiotics, diuretics, inhalation medication, prednisolone, iv fluids, iv antibiotics
Functional level | 30 days
  Measured by proxy assessment of functional level:
  * Change in amount of home care during 30 days follow-up
  * number of change of dwelling
Re-referrals to the Acute Community Health Care Service | 30 days
  Number of re-referrals to the ACHCS
Contact to the PCP ≤ 30-days | 30 days
  Number of contact to the PCP during 30 days follow-up

OTHER OUTCOMES:
The diagnostic accuracy of FLUS conducted by ACNs | 7 days
  ACNs conclusions are index test and FLUS-specialist conclusions used as reference test.

CONTACTS AND LOCATIONS:
Overall Officials: Siri A Smedemark, MD, Principal Investigator — Department of Clinical Reasearch, University of Southern Denmark; Karen Andersen-Ranberg, Prof, MD, Study Chair — Odense University Hospital
Locations (1):
- Siri Smedemark, Kolding, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smedemark SA, Laursen CB, Jarbol DE, Rosenvinge FS, Andersen-Ranberg K. Extended use of point-of-care technology versus usual care for in-home assessment by acute community nurses in older adults with signs of potential acute respiratory disease: an open-label randomised controlled trial protocol. BMC Geriatr. 2024 Feb 16;24(1):161. doi: 10.1186/s12877-024-04774-z. PMID 38365595